CLINICAL TRIAL: NCT03290287
Title: Aclidinium Bromide Post-Authorisation Safety Study to Evaluate the Risk of Cardiovascular Endpoints: Common Study Protocol
Brief Title: Aclidinium Bromide Post-Authorisation Safety Study to Evaluate the Risk of Cardiovascular Endpoints
Acronym: PASS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: RTI Health Solutions (Other)
Responsible Party: Sponsor
Other Study IDs: D6560R00004; EUPAS13616 (Registry Identifier: ENCePP)
Record Dates: First submitted 2017-08-18; First posted 2017-09-21 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — aclidinium bromide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- New users of aclidinium bromide: This nested cohort will be composed of patients aged 40 years or older who have previously been diagnosed with COPD and who are new users of aclidinium bromide (monotherapy; concomitant with formoterol not in fixed-dose combination; and aclidinium/formoterol)
  Interventions: Drug: Aclidinium bromide
- New users of other COPD medication: This nested cohort will include patients aged 40 years or older who have previously been diagnosed with COPD and who are new users of other COPD medication: tiotropium, other LAMAs, LABA, LABA/ICS and LAMA/LABA.
  Interventions: Drug: Other COPD medication

INTERVENTIONS:
Drug: Aclidinium bromide — Administered as monotherapy, concomitant with formoterol not in fixed-dose combination, or fixed-dose aclidinium/formoterol
  Groups: New users of aclidinium bromide
Drug: Other COPD medication — Users of the following COPD medications:
  Tiotropium
  Other long-acting anticholinergic (LAMAs): glycopyrronium bromide, umeclidinium
  LABA: formoterol, salmeterol, indacaterol
  LABA/ICS (LABA in fixed-dose combinations with ICS): formoterol/budesonide, formoterol/beclometasone, formoterol/mometasone, formoterol/fluticasone, salmeterol/fluticasone, and vilanterol/fluticasone.
  LAMA/LABA (approved or under regulatory review or in development): glycopyrrolate/formoterol, glycopyrronium/indacaterol, tiotropium/olodaterol, umeclidinium/vilanterol
  Groups: New users of other COPD medication

SUMMARY:
The purpose of this study is to evaluate the potential cardiovascular safety concerns and all-cause mortality described in the risk management plan for aclidinium bromide, through sequential, nested case-control studies for each endpoint of interest

DETAILED DESCRIPTION:
This is a post-authorisation safety study (PASS) of new users of aclidinium bromide, fixed dose aclidinium bromide/formoterol fumarate dihydrate, and other inhaled medications frequently used by patients with COPD

The plan is for the PASS study to be conducted on one population-based automated health database; the initial candidate database is the CRPD in the United Kingdom.

ELIGIBILITY:
Inclusion Criteria:

1. Have at least 1 year of enrolment in the electronic database. In the CPRD, only patients with permanent registration status in "up to standard" participant general practices will be included in the cohort.
2. Be aged 40 years or older.
3. Have a recorded diagnosis of COPD.
4. Have not been prescribed a study medication of interest during the 6 months before the date of the first prescription for that specific study medication.

Exclusion Criteria:

1. Patients with cancer or other serious, non-cardiovascular, life-threatening conditions or indicators of severe comorbidity will be excluded from the study cohort.
2. Subjects who will be potentially excluded are those with the following conditions recorded in the database at any time before the date of cohort entry: cancer, HIV, respiratory failure, end-stage renal disease or dialysis, organ transplantation, drug or alcohol abuse, coma, congenital abnormalities of the heart or great arteries.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in patients aged 40 years or older diagnosed with COPD initiating treatment with aclidinium bromide or other inhaled COPD treatments. Patients must have at least 1 year of enrolment in the electronic database and to have not been prescribed the study medication of interest during the 6-months before the date of the first prescription for that specific study medication. Patients with life-threatening non-cardiovascular comorbidity (e.g., malignancy, HIV infection, other) will be excluded
Sampling Method: Probability Sample
Enrollment: 26839 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence rate of mortality from all causes | From the launch of Aclidinium Bromide in the UK (October 2012) to the end of the study period (2-3 months following start of data collection [January 2017]).
  Age- and sex-standardised incidence rate per 1,000 person-years (95% CI). Potential cases will be identified by general practitioner diagnosis, hospital discharge codes and mortality data from national statistics.

SECONDARY OUTCOMES:
Incidence rate of first-ever hospitalisation for heart failure | From the launch of Aclidinium Bromide in the UK (October 2012) to the end of the study period (2-3 months following start of data collection [First semester 2017]).
  Age- and sex-standardised incidence rate per 1,000 person-years (95% CI). Potential cases will be identified by general practitioner diagnosis, hospital discharge codes and mortality data from national statistics.
Incidence rate of hospitalisation for acute myocardial infarction (fatal or non-fatal) | From the launch of Aclidinium Bromide in the UK (October 2012) to the end of the study period (2-3 months following start of data collection [First semester 2021]).
  Including community (out-of-hospital) coronary heart disease deaths. Age- and sex-standardised incidence rate per 1,000 person-years (95% CI). Potential cases will be identified by general practitioner diagnosis, hospital discharge codes and mortality data from national statistics.
Incidence rate of acute stroke (fatal or non-fatal) | From the launch of Aclidinium Bromide in the UK (October 2012) to the end of the study period (2-3 months following start of data collection [First semester 2020]).
  Including community (out-of-hospital) cerebrovascular disease deaths. Age- and sex-standardised incidence rate per 1,000 person-years (95% CI). Potential cases will be identified by general practitioner diagnosis, hospital discharge codes and mortality data from national statistics.
Incidence rate of new episodes of any type of diagnosed cardiac arrhythmia | From the launch of Aclidinium Bromide in the UK (October 2012) to the end of the study period (2-3 months following start of data collection [First semester 2022]).
  Age- and sex-standardised incidence rate per 1,000 person-years (95% CI). Potential cases will be identified by general practitioner diagnosis, hospital discharge codes and mortality data from national statistics.

OTHER OUTCOMES:
Relative risk of acute myocardial infarction, stroke, and out-of-hospital coronary heart disease or cerebrovascular death | From the launch of Aclidinium Bromide in the UK (October 2012) to the end of the study period of individual components (2-3 months following start of data collection).
  A composite endpoint of acute myocardial infarction, stroke, and out-of-hospital coronary heart disease or cerebrovascular death (if confirmed that the direction and magnitude of the risk is similar across the individual components). Potential cases will be identified by general practitioner diagnosis, hospital discharge codes and mortality data from national statistics.
Incidence rate of new episodes of atrial fibrillation or flutter | From the launch of Aclidinium Bromide in the UK (October 2012) to the end of the study period (2-3 months following start of data collection [First semester 2022]).
  Including episodes of paroxysmal (intermittent) atrial fibrillation or a new episode (first ever) or atrial fibrillation in patients without atrial fibrillation or flutter. Age- and sex-standardised incidence rate per 1,000 person-years (95% CI). Potential cases will be identified by general practitioner diagnosis, hospital discharge codes and mortality data from national statistics.
Incidence rate of new episodes of serious ventricular arrhythmias (SVA) | From the launch of Aclidinium Bromide in the UK (October 2012) to the end of the study period (2-3 months following start of data collection [First semester 2022]).
  Age- and sex-standardised incidence rate per 1,000 person-years (95% CI). Potential cases will be identified by general practitioner diagnosis, hospital discharge codes and mortality data from national statistics.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Practice Research Datalink, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No